CLINICAL TRIAL: NCT02370251
Title: Fish Oil Lipid Emulsion for the Treatment of Parenteral-Nutrition-Associated Liver Disease in Infants
Brief Title: Compassionate Use of Omegaven in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: OU Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5451
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Total Parenteral Nutrition-induced Cholestasis; Cholestasis; Short Bowel Syndrome; Gastroschisis; Intestinal Atresia; Infant, Premature, Diseases; Cholestasis of Parenteral Nutrition
Keywords: Fat Emulsions, Intravenous; Parenteral-Nutrition-Associated Liver Disease; Cholestasis; Omegaven; Fish Oil
MeSH Terms: conditions — Cholestasis; Short Bowel Syndrome; Gastroschisis; Intestinal Atresia; Infant, Premature, Diseases | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven (Experimental): Children will receive Omegaven at a maximum of 1 g/kg/day upon enrollment in this arm.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Once the direct bilirubin is 2 mg/dL or more x 2 weeks, Intralipid will be switched to Omegaven at 1 g/kg/day. The bilirubin level will be monitored to determine when resolution of cholestasis (DB <2 mg/dL) occurs.
  Other Names: Fish oil-based lipid; Omega-3-fatty acid lipid emulsion

SUMMARY:
This is a single-assignment study to evaluate whether Omegaven (IV fish oil) is effective at treating liver disease in children on long-term IV nutrition.

DETAILED DESCRIPTION:
Children up to 18 years of age, on parenteral nutrition, with a direct bilirubin level of 2 mg/dL or greater will be eligible to receive Omegaven at a maximum dose of 1 g/kg/day.

Up to 200 children will be eligible for enrollment.

Direct bilirubin levels and other labs will be monitored as well as growth parameters.

ELIGIBILITY:
Inclusion Criteria:

* Live in or temporarily relocate to Oklahoma
* Age less than 18 years, both sexes, all races
* Have a direct bilirubin level of ≥2 mg/dL for two consecutive weeks after at least 14 days of parenteral nutrition
* Received parenteral lipids at a maximum dose of 1.7 g/kg/day (24 g/kg over the two weeks prior)
* Are not currently enrolled in another lipid emulsion study

Exclusion Criteria:

* Known food allergy to fish
* Known metabolic disorder of lipid metabolism
* Active coagulopathies (active bleeding or requiring blood product treatment in the prior 48 hours)
* Medical condition likely to result in death in the next 30 days

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly D Ernst, MD, MSMI, Principal Investigator — The University of Oklahoma, Department of Pediatrics
Locations (1):
- OU Children's Hospital, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omegaven: Omegaven: Once the direct bilirubin is 2 mg/dL or more x 2 weeks, Intralipid will be switched to Omegaven at 1 g/kg/day.
Period: Overall Study
Arm/Group | Omegaven
Started | 63
Completed | 52
Not Completed | 11
Not completed — Received less than 8 days of Omegaven | 7
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Infants who required at least 8 days of Omegaven and death did not occur while on Omegaven.
Arm/Group | Omegaven
Number analyzed (Participants) | 52
Age, Customized [Mean (Inter-Quartile Range); unit: weeks]
  Birth Gestational Age | 30 [26 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52
Birth Weight (g) [Mean (Inter-Quartile Range); unit: grams] | 1410 [859 to 1768]

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Cholestasis for Subjects Who Received Omegaven
Description: To determine if Omegaven results in the resolution of cholestasis (DB <2 for 2 consecutive weeks)
Time Frame: Within the first 3 months of sole Omegaven use
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 52
Participants
  Cholestasis resolved within 3 months | 40
  Cholestasis resolved after 3 months | 10
  Cholestasis not resolved | 2

2. Secondary Outcome: Safety Issues for Infants Who Received Omegaven
Description: To determine if Omegaven results in safety issues such as increased bleeding, essential fatty acid deficiency, elevated liver function tests, increased liver and/or intestinal transplant rates, or death
Time Frame: Within the first year of use
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 52
Participants
  Baseline : INR >1.4 | 10
  End of Treatment : INR >1.4 | 7
  Baseline : Gamma-Glutamyl Transferase (GGT) >300 | 6
  End of Treatment : GGT >300 | 7
  Baseline : High-density Lipoprotein (HDL) <20 | 39
  End of Treatment : HDL <20 | 24

3. Secondary Outcome: Essential Fatty Acid Deficiency in Infants Who Received Omegaven
Description: To determine if Omegaven can resolve essential fatty acid deficiency
Time Frame: Within the first month of use
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 52
Participants
  Did not have EFAD | 14
  EFAD resolved | 27
  EFAD not resolved | 11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Omegaven
All-Cause Mortality (participants affected / at risk) | 4/52
Serious Adverse Events (participants affected / at risk) | 9/52
Other Adverse Events (participants affected / at risk) | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omegaven (N=52)
Elevated INR (Blood and lymphatic system disorders) | 4
Elevated GGT (Hepatobiliary disorders) | 5

LIMITATIONS AND CAVEATS:
This was a compassionate use study, using Omegaven as a "last resort" for infants with a direct bilirubin of at least 2 mg/dL at the time of initiation, so these infants were already at higher risk of death and hematological/hepatobiliary morbidity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02370251/Prot_SAP_000.pdf